CLINICAL TRIAL: NCT04975360
Title: Effects of a Time-delayed, Pulsatile Caffeine Formula on Sleep Inertia, Morning Cognition, Affect and Sleepiness in Healthy Volunteers
Brief Title: Delayed-release Bedtime Caffeine and Sleep Inertia Symptoms Immediately Upon Awakening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Lokman Hekim University (Other Government); Elixir Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Hans-Peter Landolt, Research Director, University of Zurich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Caff-Clock
Record Dates: First submitted 2021-02-03; First posted 2021-07-23 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Sleep Inertia; Caffeine; Placebo
Keywords: Sleep restriction; Proactive countermeasure
MeSH Terms: conditions — Idiopathic Hypersomnia | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo controlled, cross-over design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): Administration of a time-controlled, pulsatile-release caffeine formulation (160 mg caffeine) at 22:30. Participants are kept awake until 03:00 and then given a 4-hour sleep opportunity.
  Interventions: Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): Administration of a placebo formulation at 22:30. Participants are kept awake until 03:00 and then given a 4-hour sleep opportunity.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — The 160 mg caffeine pulsatile-release formulation was manufactured using a drug layering process. Caffeine and the excipients are dispersed in the coating media and then sprayed onto inert microcrystalline cellulose spheres using a fluid bed through a Wurster tube with continuous inlet air that dries the liquid in the dispersion, to obtain various layers consisting of caffeine and release-controlling polymers. The applied release-controlling polymeric system is based on methacrylate copolymers, which control the release of caffeine in pH-dependent and pH-independent manner. The release mechanism of the polymeric system is mainly driven by the swellability and permeability of the copolymers. The final micropellets are then encapsulated into hydroxypropylmethylcellulose capsules.
  Arms: Caffeine
Other: Placebo — Identical hydroxypropylmethylcellulose capsules without containing caffeine micropellets.
  Arms: Placebo

SUMMARY:
Sleep inertia (sometimes also referred to as sleep drunkenness) is a disabling state of increased sleepiness, impaired mood and reduced vigilance immediately upon awakening. Sleep inertia is highly prevalent in various neurological diseases, including neurodegenerative, affective and circadian sleep-wake rhythms disorders, as well as in frequent societal conditions such as chronic sleep restriction, jetlag and shiftwork. Reactive countermeasures against sleep inertia, i.e., strategies implemented upon wake-up, are not sufficiently effective, yet current recommendations are limited to proactive strategies, including long enough sleep at optimal times of day. These recommendations are not always easy and sometimes impossible to apply. To address this unmet medical need, the investigators developed an innovative, time-controlled, pulsatile-release formulation of 160 mg caffeine targeting an efficacious dose briefly before planned awakening.

DETAILED DESCRIPTION:
Sleep inertia is a disabling state of grogginess and impaired vigilance immediately upon awakening. The adenosine receptor antagonist, caffeine, is widely used to reduce sleep inertia symptoms, yet the initial, most severe impairments are hardly alleviated by post-awakening caffeine intake. To ameliorate this disabling state more potently, the investigators developed an innovative, delayed, pulsatile-release caffeine formulation targeting an efficacious dose briefly before planned awakening.

The investigators comprehensively test this formulation in two placebo-controlled, double-blind, cross-over studies. First, the investigators establish the in vivo caffeine release profile in young men. Subsequently, they investigate the formulation's ability to improve sleep inertia in sleep-restricted volunteers. Following oral administration of 160 mg caffeine at habitual bedtime [22:30], the investigators keep the participants awake until 03:00, to increase sleep inertia symptoms upon scheduled awakening [at 07:00]. Immediately upon awakening, the investigators quantify subjective state, psychomotor vigilance, cognitive performance, and the cortisol awakening response. They also record polysomnography during nocturnal sleep and a 1-hour nap opportunity at 08:00.

ELIGIBILITY:
Inclusion Criteria:

* male sex in order to avoid the potential impact of menstrual cycle on sleep physiology or HPA axis activity,
* age within the range of 18 to 34 years,
* a body-mass-index below 25,
* an Epworth Sleepiness Score (ESS) below 10,
* habitual sleep onset latency below 20 minutes,
* regular sleep-wake rhythm with bedtime between 11 pm and 1 am,
* absence of any somatic or psychiatric disorders,
* no acute or chronic medication intake,
* non-smoking,
* no history of drug abuse (lifetime use > 5 occasions, except occasional cannabis use)
* caffeine consumption of less than 4 units per day (coffee, tea, chocolate, cola, energy drinks)

Exclusion Criteria:

- Failure to meet inclusion criteria

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Acute Sleep Inertia Questionnaire | At 07:00 hours after caffeine and placebo administration
  Modified questionnaire to assess subjective ratings of sleep inertia on physiological, emotional, cognitive and behavioral levels.

SECONDARY OUTCOMES:
Polysomnographic recording of nocturnal sleep | Between 03:00-07:00 hours after caffeine and placebo administration
  All-night polysomnographic recordings of nocturnal sleep: electrical bio-signals include simultaneous, standardized recordings of brain waves (electroencephalogram), muscle tone on the chin (electromyogram), and slow and rapid eye movements (electrooculogram). The information will be aggregated for visual scoring of sleep stages according to standardized criteria specified by the American Academy of Sleep Medicine.
Caffeine Effects Questionnaire | Between 07:15-08:00 hours after caffeine and placebo administration
  Acute questionnaire to assess caffeine-related subjective effects.
Positive and Negative Affect Schedule | Between 07:00-08:15 hours after caffeine and placebo administration
  Questionnaire
Psychomotor vigilance task | Between 07:15-07:30 hours after caffeine and placebo administration
  Reaction-time task
N-back task | Between 07:30-07:40 hours after caffeine and placebo administration
  Working memory and brain executive function task
d2 attention task | Between 07:40-07:45 hours after caffeine and placebo administration
  Focused attention task
Cortisol awakening response | Between 07:00-08:00 hours after caffeine and placebo administration
  Physiological awakening response to address HPA-axis function
Polysomnographic recording of morning nap opportunity | Between 08:00-09:00 hours after caffeine and placebo administration
  Polysomnographic recordings of sleep during one-hour nap opportunity: electrical bio-signals include simultaneous, standardized recordings of brain waves (electroencephalogram), muscle tone on the chin (electromyogram), and slow and rapid eye movements (electrooculogram). The information will be aggregated for visual scoring of sleep stages according to standardized criteria specified by the American Academy of Sleep Medicine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dornbierer DA, Yerlikaya F, Wespi R, Boxler MI, Voegel CD, Schnider L, Arslan A, Baur DM, Baumgartner MR, Binz TM, Kraemer T, Landolt HP. A novel bedtime pulsatile-release caffeine formula ameliorates sleep inertia symptoms immediately upon awakening. Sci Rep. 2021 Oct 5;11(1):19734. doi: 10.1038/s41598-021-98376-z. PMID 34611208